CLINICAL TRIAL: NCT07380022
Title: Acceptability, Adherence, and Impact on the Bioavailability of Iron and Zinc of the Dietary Supplements Goodphyte IB Defense and Goodphyte Immunity in Adults With Chronic Diseases.
Acronym: PHYTASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vaios Svolos, Dietitian, Postdoctoral Researcher, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 92/25.6.2025
Record Dates: First submitted 2025-12-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: IBD; Hypertension (HTN); Multiple Sclerosis; Anemia; Colitis Ulcerative
Keywords: ACCEPTABILITY; DIETARY SUPPLEMENT; PHYTASE
MeSH Terms: conditions — Hypertension; Multiple Sclerosis; Anemia; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement intervention Goodphyte IB Defense (Other): 50 Participants will receive dietary supplement Goodphyte IB Defense
  Interventions: Dietary Supplement: Dietary supplement intervention Goodphyte IB Defense
- Dietary supplement intervention Goodphyte Immunity (Other): 50 Participants will receive dietary supplement Goodphyte Immunity
  Interventions: Dietary Supplement: Dietary supplement intervention Goodphyte Immunity

INTERVENTIONS:
Dietary Supplement: Dietary supplement intervention Goodphyte IB Defense — Participants will receive orally Goodphyte IB Defense at a dose of four capsules per day for a duration of two weeks.
  Arms: Dietary supplement intervention Goodphyte IB Defense
Dietary Supplement: Dietary supplement intervention Goodphyte Immunity — Participants will receive orally Goodphyte IB Immunity at a dose of four capsules per day for a duration of two weeks.
  Arms: Dietary supplement intervention Goodphyte Immunity

SUMMARY:
The primary objective of the present postdoctoral research is to evaluate the acceptability and adherence of two dietary supplements containing microbial phytase, Goodphyte IB Defense and Goodphyte Immunity, in adult individuals with chronic diseases, namely Idiopathic Inflammatory Bowel Diseases (IIBD)-that is, Crohn's disease (CD) or Ulcerative Colitis (UC)-Arterial Hypertension (AH), Anemia (AN), or Multiple Sclerosis (MS).

Secondarily, this study will investigate potential changes in iron and zinc absorption following phytase supplementation in these individuals and, consequently, possible changes in their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease: Patients in remission, with a stable type of pharmacological treatment over the past 3 months and a stable dosage during the last month.
* Ulcerative colitis: Patients in remission, with a stable type of pharmacological treatment over the past 3 months and a stable dosage during the last month.
* Hypertension: Patients with systolic blood pressure of 130-139 mmHg or diastolic blood pressure of 80-89 mmHg, who maintain blood pressure within these ranges through lifestyle modifications, without active symptoms (e.g., headaches, dizziness), and not receiving antihypertensive medication.
* Anemia: Patients with hemoglobin <12 g/dL, serum iron <40 μg/dL, and ferritin <15 ng/mL for women, and hemoglobin <13 g/dL, serum iron <40 μg/dL, and ferritin <30 ng/mL for men. Absence of severe clinical consequences. Presence of fatigue, weakness, or dizziness, which is usually manageable.
* Multiple sclerosis: Patients in remission, with a stable type of pharmacological treatment over the past 3 months and a stable dosage during the last month.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Current use of antibiotics or antibiotic use within the past month
* Current use of other probiotic, prebiotic, or synbiotic supplements
* Current use of iron and/or zinc supplements
* Change in the type of therapeutic regimen (pharmacotherapy) within the past three months
* Change in the dosage of the therapeutic regimen (pharmacotherapy) within the past month
* Renal or hepatic disease
* Inability to provide informed consent (including individuals <18 years of age)
* Insufficient understanding of the Greek language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Acceptability of two dietary supplements containing microbial phytase, Goodphyte IB Defense and Goodphyte Immunity using an acceptability questionnaire | 2 weeks (immediately after completion of the 2-week intervention)
  Acceptability will be measured using an acceptability questionnaire completed at the end of the intervention. The questionnaire will include items assessing ease of intake, difficulties in integrating the supplement into daily routines, perceived safety, overall study experience, and intention to continue product use. Responses will be recorded using a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), allowing quantitative analysis.
Adherence to the Intervention | From enrollment to the end of treatment at 2 weeks
  Adherence will be assessed by recording the number of days participants consumed the supplement and the quantity consumed during the intervention period. Daily adherence will be documented using a self-reported compliance form. Participant completion and withdrawal rates will be recorded, and reasons for withdrawal will be analyzed when available.

SECONDARY OUTCOMES:
Changes in serum iron levels (μg/dL) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  The effect of supplementation with Goodphyte IB Defense and Goodphyte Immunity on iron status will be evaluated. Blood samples will be collected before and after the intervention to measure serum iron. All laboratory analyses will be performed using standardized and validated methods.
Changes in serum zinc levels (μg/dL) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  The effect of supplementation with Goodphyte IB Defense and Goodphyte Immunity on zinc status will be evaluated. Blood samples will be collected before and after the intervention to measure serum zinc. All laboratory analyses will be performed using standardized and validated methods.
Changes in ferritin (ng/mL) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  The effect of supplementation with Goodphyte IB Defense and Goodphyte Immunity on inflammatory markers will be evaluated. Blood samples will be collected before and after the intervention to measure ferritin. All laboratory analyses will be performed using standardized and validated methods.
Changes in C-reactive protein (CRP) (mg/L) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  The effect of supplementation with Goodphyte IB Defense and Goodphyte Immunity on inflammatory markers will be evaluated. Blood samples will be collected before and after the intervention to measure C-reactive protein (CRP). All laboratory analyses will be performed using standardized and validated methods.
Changes in fecal calprotectin (µg/g) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  In participants with Inflammatory Bowel Disease (IBD), fecal calprotectin will be measured as a non-invasive marker of intestinal inflammation. Stool samples will be collected before and after the intervention. All laboratory analyses will be performed using standardized and validated methods.
Changes in Erythrocyte Sedimentation Rate (ESR) (mm) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  The effect of supplementation with Goodphyte IB Defense and Goodphyte Immunity on inflammatory markers will be evaluated. Blood samples will be collected before and after the intervention to measure Erythrocyte Sedimentation Rate (ESR). All laboratory analyses will be performed using standardized and validated methods.
Changes in Quality of Life (QoL) using WHOQOL-BREF questionnaire | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Quality of Life (QoL) will be assessed using internationally recognized questionnaire for the evaluation of participants' subjective well-being, such as WHOQOL-BREF: The World Health Organization Quality of Life-Abbreviated version. Domain scores will be calculated and transformed to a 0-100 scale according to World Health Organization guidelines, with higher scores indicating better quality of life.
Changes in Quality of Life (QoL) using EQ-5D-5L questionnaire | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Quality of Life (QoL) will be assessed using internationally recognized questionnaire for the evaluation of participants' subjective well-being, such as EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L). The EQ-5D-5L index score will be calculated using the validated country-specific value set, converting health states into a single index value ranging from 0 to 1, where higher values indicate better health-related quality of life.
Changes in fatigue levels using the Chalder Fatigue Scale (CFQ) questionnaire | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Participants will complete the Chalder Fatigue Scale (CFQ) questionnaire, which consists of 11 Likert-scale questions designed to distinguish between physical and mental fatigue. Responses will be scored using the Likert method (0-3), yielding a total fatigue score ranging from 0 to 33, with higher scores indicating greater fatigue severity.
Body Mass Index (BMI) using measured body weight and height (kg/m²) | Baseline (Day 0) and 2 weeks (immediately after completion of the 2-week intervention)
  Body Mass Index (BMI) will be assessed as a measure of body composition. BMI will be calculated using measured body weight and height (kg/m²) at baseline, during the intervention, and at the end of the intervention to evaluate changes over time.
Harvey-Bradshaw Index (HBI) Score | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Self-reported disease activity in patients with Crohn's disease will be assessed using the Harvey-Bradshaw Index (HBI), summing points from general well-being, abdominal pain, liquid stools, abdominal mass, and complications. Scores typically indicate: <5 (remission), 5-7 (mild), 8-16 (moderate), and >16 (severe) activity.
Mayo Score for Ulcerative Colitis | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Self-reported disease activity in patients with ulcerative colitis will be assessed using the Mayo Score, a 0-12 point system assessing disease severity by combining patient symptoms (stool frequency, rectal bleeding) with endoscopic findings (mucosal appearance) and a physician's global assessment, with higher scores indicating more severe inflammation.
Inflammatory Bowel Disease Disk (IBD-Disk) Score | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Patient-reported symptom severity and disease-related burden in ulcerative colitis and Crohn's disease will be assessed using the Inflammatory Bowel Disease Disk (IBD-Disk) tool. It is a 10-item, visual, self-administered tool. Patients rate 10 key areas (like abdominal pain, energy, sleep, emotions) on a 0-10 scale, resulting in a total score from 0 to 100, where higher scores indicate greater disability.
Multiple Sclerosis Impact Scale (MSIS-29) Score | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Self-reported physical and psychological impact of multiple sclerosis will be assessed using the Multiple Sclerosis Impact Scale (MSIS-29). The scores will be summed and converted to a 0-100 scale for each domain, with 100 being the worst.
Modified Fatigue Impact Scale (MFIS) Score | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Fatigue severity and its impact on daily functioning in patients with multiple sclerosis will be assessed using the Modified Fatigue Impact Scale (MFIS). It reflects how fatigue affects daily life, with a total range of 0-84, where higher scores mean greater impact, broken into physical (0-36), cognitive (0-40), and psychosocial (0-8) subscales.
Hypertension-Related Symptom Score | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Self-reported hypertension-related symptoms, including dizziness and headache, assessed using a weekly symptom questionnaire. Symptom severity will be evaluated at baseline, during the intervention, and at the end of the intervention.
Anemia-Related Symptom Score | Day 0 (baseline), Day 7 (mid-intervention) and Day 14 (immediately after completion of the 2-week intervention)
  Self-reported anemia-related symptoms, including fatigue, shortness of breath, and weakness, assessed using a weekly symptom questionnaire. Assessments will be conducted at baseline, during the intervention, and at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: ODYSSEAS ANDROUTSOS, Study Director — School of Physical Education, Sport Science and Dietetics
Locations (1):
- School of Physical Education, Sport Science and Dietetics, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No